CLINICAL TRIAL: NCT02372773
Title: Longitudinal Evaluation of Familial Frontotemporal Dementia Subjects
Acronym: LEFFTDS
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Bradley Boeve, Professor of Neurology, Mayo Clinic
Other Study IDs: 14-007532; U01AG045390 (NIH)
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Familial Frontotemporal Dementia
Keywords: Frontotemporal Dementia; MAPT; PGRN; C9ORF72
MeSH Terms: conditions — Frontotemporal Dementia; Frontotemporal Dementia With Motor Neuron Disease

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood - DNA, Plasma, Serum, Peripheral blood mononuclear cells, RNA, Cerebrospinal Fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Frontotemporal Dementia - MAPT: Frontotemporal Dementia with microtubule associated protein tau (MAPT) mutation
- Frontotemporal Dementia - PGRN: Frontotemporal Dementia with progranulin (PGRN; also known as granulin or GRN) mutation
- Frontotemporal Dementia - C9OR72: Frontotemporal Dementia with chromosome 9 open reading frame 72 (C9ORF72) mutation.
- Control: Member of family with a known mutation in one of the three major FTD related genes: MAPT, PGRN, and C9ORF72.

SUMMARY:
This study is being done to learn more about normal thinking and behavior, mild thinking and behavior problems, Frontotemporal Dementia and other forms of dementia in families in which one or more relatives have a mutation associated with Frontotemporal Dementia.

DETAILED DESCRIPTION:
This multicenter study will enroll 300 members of familial Frontotemporal Dementia (FTD) families across 8 experienced FTD research centers with a known mutation in MAPT, PGRN, or C9ORF72 (100 mutation carriers with mild dementia or minimally symptomatic yet non-demented, 100 asymptomatic mutation carriers, and 100 clinically normal relatives who are non-mutation carriers) to obtain annual assessments including T1-MRI, FLAIR, diffusion tensor imaging (DTI), ASL perfusion (ASLp), intrinsic connectivity functional MRI (icfMRI), MR spectroscopy (MRS), CSF, blood, and behavioral, neuropsychological and functional assessment, for a total of three assessments per participant.

A primary goal of this study is to identify the most robust and reliable methods to track disease progression in familial FTD so that disease-modifying therapeutic trials can be designed appropriately.

ELIGIBILITY:
Inclusion Criteria:

1. Must be a member of family with a known mutation in one of the three major FTLD related genes: MAPT, PGRN, or C9ORF72.
2. At least 18 years of age.
3. The predominant phenotype in the kindred must be cognitive/behavioral (ie, kindreds in whom parkinsonism or ALS is the predominant clinical phenotype among affected relatives may be excluded)
4. Have a reliable informant who personally speaks with or sees that subject at least weekly.
5. Subject is sufficiently fluent in English to complete all measures
6. Subject must be willing and able to consent to the protocol and undergo yearly evaluations over 3 years.
7. Subject must be willing and able to undergo neuropsychological testing (at least at baseline visit).
8. Subject must have no contraindication to MRI imaging.

Exclusion Criteria

1. Known presence of a structural brain lesion (e.g. tumor, cortical infarct).
2. Presence of another neurologic disorder which could impact findings (eg, multiple sclerosis).
3. Subject is unwilling to return for follow-up yearly, undergo neuropsychological testing and MR imaging.
4. Subject has no reliable informant.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Have a mutation, or be a relative of an individual with a mutation, in one of the three most common genes associated with Frontotemporal Dementia - microtubule associated protein tau (MAPT), progranulin (PGRN; also known as granulin or GRN), or chromosome 9 open reading frame 72 (C9ORF72).
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2015-04; Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Rate of decline in traditional measures of clinical (neuropsychological and behavioral composites) function and cortical volume on structural MRI in the symptomatic phase of familial FTD | 5 years
  neuropsychological, clinical/behavioral, neuroimaging measures

SECONDARY OUTCOMES:
Rate of decline in traditional measures of clinical (neuropsychological and behavioral composites) function and cortical volume on structural MRI in the asymptomatic phase of familial FTD | 5 years
  neuropsychological, clinical/behavioral, neuroimaging measures
Value of novel imaging and clinical measures for characterizing asymptomatic familial FTD subjects, and factors predicting clinical rates of progression in each group. | 5 years
  neuropsychological, clinical/behavioral, neuroimaging measures
Genetic and biofluid factors that modify rates of clinical and neuroimaging decline in the asymptomatic and symptomatic phases of familial FTD. | 5 years
  genetic and biolfuid factors

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Boeve, MD, Principal Investigator — Mayo Clinic; Howard Rosen, MD, Principal Investigator — University of California, San Francisco
Locations (8):
- United States (7):
  - University of California, San Francisco, Memory and Aging Center, Department of Neurology, San Francisco, California
  - Mayo Clinic Florida, Jacksonville, Florida
  - Harvard University, Charlestown, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Univerisity of Pennsylvania, Philadelphia, Pennsylvania
- University of British Columbia, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data can be shared following a formal request and approval by the executive committee overseeing the protocol.
Supporting Information: Study Protocol
Time Frame: De-identified data is available throughout course of the protocol.
Access Criteria: De-identified data can be shared following a formal request and approval by the executive committee overseeing the protocol. Requests can be made be completing the data request form at this site: https://ucsf.co1.qualtrics.com/jfe/form/SV_e4BBGMiXV7HRTg1
URL: https://ucsf.co1.qualtrics.com/jfe/form/SV_e4BBGMiXV7HRTg1

REFERENCES:
- [Result] Gentry MT, Lapid MI, Syrjanen J, Calvert K, Hughes S, Brushaber D, Kremers W, Bove J, Brannelly P, Coppola G, Dheel C, Dickerson B, Dickinson S, Faber K, Fields J, Fong J, Foroud T, Forsberg L, Gavrilova R, Gearhart D, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford N, Grossman M, Haley D, Heuer H, Hsiung GY, Huey E, Irwin D, Jones D, Jones L, Kantarci K, Karydas A, Knopman D, Kornak J, Kramer J, Kukull W, Lucente D, Lungu C, Mackenzie I, Manoochehri M, McGinnis S, Miller B, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin K, Rascovsky K, Sengdy P, Shaw L, Tatton N, Taylor J, Toga A, Trojanowski J, Weintraub S, Wong B, Wszolek Z, Boeve BF, Boxer A, Rosen H; LEFFTDS Consortium. Quality of life and caregiver burden in familial frontotemporal lobar degeneration: Analyses of symptomatic and asymptomatic individuals within the LEFFTDS cohort. Alzheimers Dement. 2020 Aug;16(8):1115-1124. doi: 10.1002/alz.12095. Epub 2020 Jul 13. PMID 32656921
- [Result] Thijssen EH, La Joie R, Wolf A, Strom A, Wang P, Iaccarino L, Bourakova V, Cobigo Y, Heuer H, Spina S, VandeVrede L, Chai X, Proctor NK, Airey DC, Shcherbinin S, Duggan Evans C, Sims JR, Zetterberg H, Blennow K, Karydas AM, Teunissen CE, Kramer JH, Grinberg LT, Seeley WW, Rosen H, Boeve BF, Miller BL, Rabinovici GD, Dage JL, Rojas JC, Boxer AL; Advancing Research and Treatment for Frontotemporal Lobar Degeneration (ARTFL) investigators. Diagnostic value of plasma phosphorylated tau181 in Alzheimer's disease and frontotemporal lobar degeneration. Nat Med. 2020 Mar;26(3):387-397. doi: 10.1038/s41591-020-0762-2. Epub 2020 Mar 2. PMID 32123386
- [Result] Chen Q, Boeve BF, Senjem M, Tosakulwong N, Lesnick T, Brushaber D, Dheel C, Fields J, Forsberg L, Gavrilova R, Gearhart D, Graff-Radford J, Graff-Radford N, Jack CR Jr, Jones D, Knopman D, Kremers WK, Lapid M, Rademakers R, Ramos EM, Syrjanen J, Boxer AL, Rosen H, Wszolek ZK, Kantarci K. Trajectory of lobar atrophy in asymptomatic and symptomatic GRN mutation carriers: a longitudinal MRI study. Neurobiol Aging. 2020 Apr;88:42-50. doi: 10.1016/j.neurobiolaging.2019.12.004. Epub 2019 Dec 12. PMID 31918955
- [Result] Staffaroni AM, Bajorek L, Casaletto KB, Cobigo Y, Goh SM, Wolf A, Heuer HW, Elahi FM, Ljubenkov PA, Dever R, Kornak J, Appleby B, Bove J, Bordelon Y, Brannelly P, Brushaber D, Caso C, Coppola G, Dheel C, Dickerson BC, Dickinson S, Dominguez S, Domoto-Reilly K, Faber K, Ferrall J, Fields JA, Fishman A, Fong J, Foroud T, Forsberg LK, Gavrilova R, Gearhart D, Ghazanfari B, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford N, Grant I, Grossman M, Haley D, Hsiung GY, Huey ED, Irwin DJ, Jones DT, Jones L, Kantarci K, Karydas A, Kaufer DI, Kerwin DR, Knopman DS, Kraft R, Kremers WK, Kukull WA, Litvan I, Lucente D, Lungu C, Mackenzie IR, Maldonado M, Manoochehri M, McGinnis SM, McKinley E, Mendez MF, Miller BL, Multani N, Onyike C, Padmanabhan J, Pantelyat A, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin KP, Rascovsky K, Roberson ED, Rogalski E, Sengdy P, Shaw LM, Syrjanen J, Tartaglia MC, Tatton N, Taylor J, Toga A, Trojanowski JQ, Weintraub S, Wang P, Wong B, Wszolek Z, Boxer AL, Boeve BF, Kramer JH, Rosen HJ; ARTFL/LEFFTDS consortium. Assessment of executive function declines in presymptomatic and mildly symptomatic familial frontotemporal dementia: NIH-EXAMINER as a potential clinical trial endpoint. Alzheimers Dement. 2020 Jan;16(1):11-21. doi: 10.1016/j.jalz.2019.01.012. PMID 31914230
- [Result] Heuer HW, Wang P, Rascovsky K, Wolf A, Appleby B, Bove J, Bordelon Y, Brannelly P, Brushaber DE, Caso C, Coppola G, Dickerson B, Dickinson S, Domoto-Reilly K, Faber K, Ferrall J, Fields J, Fishman A, Fong J, Foroud T, Forsberg LK, Gearhart D, Ghazanfari B, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford N, Grant I, Grossman M, Haley D, Hsiung GY, Huey E, Irwin D, Jones D, Kantarci K, Karydas A, Kaufer D, Kerwin D, Knopman D, Kornak J, Kramer JH, Kraft R, Kremers WK, Kukull W, Litvan I, Ljubenkov P, Mackenzie IR, Maldonado M, Manoochehri M, McGinnis S, McKinley E, Mendez MF, Miller BL, Onyike C, Pantelyat A, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin KP, Roberson ED, Rogalski E, Sengdy P, Shaw L, Syrjanen J, Tartaglia MC, Tatton N, Taylor J, Toga A, Trojanowski J, Weintraub S, Wong B, Wszolek Z, Boeve BF, Rosen HJ, Boxer AL; ARTFL and LEFFTDS consortia. Comparison of sporadic and familial behavioral variant frontotemporal dementia (FTD) in a North American cohort. Alzheimers Dement. 2020 Jan;16(1):60-70. doi: 10.1002/alz.12046. PMID 31914226
- [Result] Rosen HJ, Boeve BF, Boxer AL. Tracking disease progression in familial and sporadic frontotemporal lobar degeneration: Recent findings from ARTFL and LEFFTDS. Alzheimers Dement. 2020 Jan;16(1):71-78. doi: 10.1002/alz.12004. PMID 31914219
- [Result] Miyagawa T, Brushaber D, Syrjanen J, Kremers W, Fields J, Forsberg LK, Heuer HW, Knopman D, Kornak J, Boxer A, Rosen HJ, Boeve BF, Appleby B, Bordelon Y, Bove J, Brannelly P, Caso C, Coppola G, Dever R, Dheel C, Dickerson B, Dickinson S, Dominguez S, Domoto-Reilly K, Faber K, Ferrell J, Fishman A, Fong J, Foroud T, Gavrilova R, Gearhart D, Ghazanfari B, Ghoshal N, Goldman JS, Graff-Radford J, Graff-Radford N, Grant I, Grossman M, Haley D, Hsiung R, Huey E, Irwin D, Jones D, Jones L, Kantarci K, Karydas A, Kaufer D, Kerwin D, Kraft R, Kramer J, Kukull W, Litvan I, Lucente D, Lungu C, Mackenzie I, Maldonado M, Manoochehri M, McGinnis S, McKinley E, Mendez MF, Miller B, Multani N, Onyike C, Padmanabhan J, Pantelyat A, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin K, Rascovsky K, Roberson ED, Rogalski E, Sengdy P, Shaw L, Tartaglia MC, Tatton N, Taylor J, Toga A, Trojanowski JQ, Wang P, Weintraub S, Wong B, Wszolek Z. Utility of the global CDR(R) plus NACC FTLD rating and development of scoring rules: Data from the ARTFL/LEFFTDS Consortium. Alzheimers Dement. 2020 Jan;16(1):106-117. doi: 10.1002/alz.12033. PMID 31914218
- [Result] Ramos EM, Dokuru DR, Van Berlo V, Wojta K, Wang Q, Huang AY, Deverasetty S, Qin Y, van Blitterswijk M, Jackson J, Appleby B, Bordelon Y, Brannelly P, Brushaber DE, Dickerson B, Dickinson S, Domoto-Reilly K, Faber K, Fields J, Fong J, Foroud T, Forsberg LK, Gavrilova R, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford N, Grant I, Grossman M, Heuer HW, Hsiung GR, Huey E, Irwin D, Kantarci K, Karydas A, Kaufer D, Kerwin D, Knopman D, Kornak J, Kramer JH, Kremers W, Kukull W, Litvan I, Ljubenkov P, Lungu C, Mackenzie I, Mendez MF, Miller BL, Onyike C, Pantelyat A, Pearlman R, Petrucelli L, Potter M, Rankin KP, Rascovsky K, Roberson ED, Rogalski E, Shaw L, Syrjanen J, Tartaglia MC, Tatton N, Taylor J, Toga A, Trojanowski JQ, Weintraub S, Wong B, Wszolek Z, Rademakers R, Boeve BF, Rosen HJ, Boxer AL; ARTFL/LEFFTDS consortium; Coppola G. Genetic screening of a large series of North American sporadic and familial frontotemporal dementia cases. Alzheimers Dement. 2020 Jan;16(1):118-130. doi: 10.1002/alz.12011. PMID 31914217
- [Result] Moore KM, Nicholas J, Grossman M, McMillan CT, Irwin DJ, Massimo L, Van Deerlin VM, Warren JD, Fox NC, Rossor MN, Mead S, Bocchetta M, Boeve BF, Knopman DS, Graff-Radford NR, Forsberg LK, Rademakers R, Wszolek ZK, van Swieten JC, Jiskoot LC, Meeter LH, Dopper EG, Papma JM, Snowden JS, Saxon J, Jones M, Pickering-Brown S, Le Ber I, Camuzat A, Brice A, Caroppo P, Ghidoni R, Pievani M, Benussi L, Binetti G, Dickerson BC, Lucente D, Krivensky S, Graff C, Oijerstedt L, Fallstrom M, Thonberg H, Ghoshal N, Morris JC, Borroni B, Benussi A, Padovani A, Galimberti D, Scarpini E, Fumagalli GG, Mackenzie IR, Hsiung GR, Sengdy P, Boxer AL, Rosen H, Taylor JB, Synofzik M, Wilke C, Sulzer P, Hodges JR, Halliday G, Kwok J, Sanchez-Valle R, Llado A, Borrego-Ecija S, Santana I, Almeida MR, Tabuas-Pereira M, Moreno F, Barandiaran M, Indakoetxea B, Levin J, Danek A, Rowe JB, Cope TE, Otto M, Anderl-Straub S, de Mendonca A, Maruta C, Masellis M, Black SE, Couratier P, Lautrette G, Huey ED, Sorbi S, Nacmias B, Laforce R Jr, Tremblay ML, Vandenberghe R, Damme PV, Rogalski EJ, Weintraub S, Gerhard A, Onyike CU, Ducharme S, Papageorgiou SG, Ng ASL, Brodtmann A, Finger E, Guerreiro R, Bras J, Rohrer JD; FTD Prevention Initiative. Age at symptom onset and death and disease duration in genetic frontotemporal dementia: an international retrospective cohort study. Lancet Neurol. 2020 Feb;19(2):145-156. doi: 10.1016/S1474-4422(19)30394-1. Epub 2019 Dec 3. PMID 31810826
- [Result] Olney NT, Ong E, Goh SM, Bajorek L, Dever R, Staffaroni AM, Cobigo Y, Bock M, Chiang K, Ljubenkov P, Kornak J, Heuer HW, Wang P, Rascovsky K, Wolf A, Appleby B, Bove J, Bordelon Y, Brannelly P, Brushaber D, Caso C, Coppola G, Dickerson BC, Dickinson S, Domoto-Reilly K, Faber K, Ferrall J, Fields J, Fishman A, Fong J, Foroud T, Forsberg LK, Gearhart DJ, Ghazanfari B, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford NR, Grant I, Grossman M, Haley D, Hsiung G, Huey ED, Irwin DJ, Jones DT, Kantarci K, Karydas AM, Kaufer D, Kerwin D, Knopman DS, Kramer JH, Kraft R, Kremers W, Kukull W, Lapid MI, Litvan I, Mackenzie IR, Maldonado M, Manoochehri M, McGinnis SM, McKinley EC, Mendez MF, Miller BL, Onyike C, Pantelyat A, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin KP, Roberson ED, Rogalski E, Sengdy P, Shaw LM, Syrjanen J, Tartaglia MC, Tatton N, Taylor J, Toga A, Trojanowski JQ, Weintraub S, Wong B, Wszolek Z, Boxer AL, Boeve BF, Rosen HJ; ARTFL and LEFFTDS consortia. Clinical and volumetric changes with increasing functional impairment in familial frontotemporal lobar degeneration. Alzheimers Dement. 2020 Jan;16(1):49-59. doi: 10.1016/j.jalz.2019.08.196. Epub 2020 Jan 6. PMID 31784375
- [Result] Boxer AL, Gold M, Feldman H, Boeve BF, Dickinson SL, Fillit H, Ho C, Paul R, Pearlman R, Sutherland M, Verma A, Arneric SP, Alexander BM, Dickerson BC, Dorsey ER, Grossman M, Huey ED, Irizarry MC, Marks WJ, Masellis M, McFarland F, Niehoff D, Onyike CU, Paganoni S, Panzara MA, Rockwood K, Rohrer JD, Rosen H, Schuck RN, Soares HD, Tatton N. New directions in clinical trials for frontotemporal lobar degeneration: Methods and outcome measures. Alzheimers Dement. 2020 Jan;16(1):131-143. doi: 10.1016/j.jalz.2019.06.4956. Epub 2020 Jan 6. PMID 31668596
- [Result] Chen Q, Boeve BF, Schwarz CG, Reid R, Tosakulwong N, Lesnick TG, Bove J, Brannelly P, Brushaber D, Coppola G, Dheel C, Dickerson BC, Dickinson S, Faber K, Fields J, Fong J, Foroud T, Forsberg L, Gavrilova RH, Gearhart D, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford NR, Grossman M, Haley D, Heuer HW, Hsiung GR, Huey E, Irwin DJ, Jack CR, Jones DT, Jones L, Karydas AM, Knopman DS, Kornak J, Kramer J, Kremers W, Kukull WA, Lapid M, Lucente D, Lungu C, Mackenzie IRA, Manoochehri M, McGinnis S, Miller BL, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin KP, Rascovsky K, Sengdy P, Shaw L, Syrjanen J, Tatton N, Taylor J, Toga AW, Trojanowski J, Weintraub S, Wong B, Boxer AL, Rosen H, Wszolek Z, Kantarci K; LEFFTDS Consortium. Tracking white matter degeneration in asymptomatic and symptomatic MAPT mutation carriers. Neurobiol Aging. 2019 Nov;83:54-62. doi: 10.1016/j.neurobiolaging.2019.08.011. Epub 2019 Aug 15. PMID 31585367
- [Result] Chen Q, Boeve BF, Senjem M, Tosakulwong N, Lesnick TG, Brushaber D, Dheel C, Fields J, Forsberg L, Gavrilova R, Gearhart D, Graff-Radford J, Graff-Radford NR, Jack CR Jr, Jones DT, Knopman DS, Kremers WK, Lapid M, Rademakers R, Syrjanen J, Boxer AL, Rosen H, Wszolek ZK, Kantarci K; LEFFTDS Consortium. Rates of lobar atrophy in asymptomatic MAPT mutation carriers. Alzheimers Dement (N Y). 2019 Jul 30;5:338-346. doi: 10.1016/j.trci.2019.05.010. eCollection 2019. PMID 31388560
- [Result] Chen Q, Boeve BF, Tosakulwong N, Lesnick T, Brushaber D, Dheel C, Fields J, Forsberg L, Gavrilova R, Gearhart D, Haley D, Gunter JL, Graff-Radford J, Jones D, Knopman D, Graff-Radford N, Kraft R, Lapid M, Rademakers R, Syrjanen J, Wszolek ZK, Rosen H, Boxer AL, Kantarci K. Frontal lobe 1H MR spectroscopy in asymptomatic and symptomatic MAPT mutation carriers. Neurology. 2019 Aug 20;93(8):e758-e765. doi: 10.1212/WNL.0000000000007961. Epub 2019 Jul 17. PMID 31315971
- [Result] Staffaroni AM, Cobigo Y, Goh SM, Kornak J, Bajorek L, Chiang K, Appleby B, Bove J, Bordelon Y, Brannelly P, Brushaber D, Caso C, Coppola G, Dever R, Dheel C, Dickerson BC, Dickinson S, Dominguez S, Domoto-Reilly K, Faber K, Ferrall J, Fields JA, Fishman A, Fong J, Foroud T, Forsberg LK, Gavrilova R, Gearhart D, Ghazanfari B, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford N, Grant I, Grossman M, Haley D, Heuer HW, Hsiung GY, Huey ED, Irwin DJ, Jones DT, Jones L, Kantarci K, Karydas A, Kaufer DI, Kerwin DR, Knopman DS, Kraft R, Kramer JH, Kremers WK, Kukull WA, Litvan I, Ljubenkov PA, Lucente D, Lungu C, Mackenzie IR, Maldonado M, Manoochehri M, McGinnis SM, McKinley E, Mendez MF, Miller BL, Multani N, Onyike C, Padmanabhan J, Pantelyat A, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin KP, Rascovsky K, Roberson ED, Rogalski E, Sengdy P, Shaw LM, Syrjanen J, Tartaglia MC, Tatton N, Taylor J, Toga A, Trojanowski JQ, Weintraub S, Wang P, Wong B, Wszolek Z, Boxer AL, Boeve BF, Rosen HJ; ARTFL/LEFFTDS consortium. Individualized atrophy scores predict dementia onset in familial frontotemporal lobar degeneration. Alzheimers Dement. 2020 Jan;16(1):37-48. doi: 10.1016/j.jalz.2019.04.007. Epub 2020 Jan 6. PMID 31272932
- [Result] Chen Q, Boeve BF, Tosakulwong N, Lesnick T, Brushaber D, Dheel C, Fields J, Forsberg L, Gavrilova R, Gearhart D, Haley D, Gunter JL, Graff-Radford J, Jones D, Knopman D, Graff-Radford N, Kraft R, Lapid M, Rademakers R, Wszolek ZK, Rosen H, Boxer AL, Kantarci K. Brain MR Spectroscopy Changes Precede Frontotemporal Lobar Degeneration Phenoconversion in Mapt Mutation Carriers. J Neuroimaging. 2019 Sep;29(5):624-629. doi: 10.1111/jon.12642. Epub 2019 Jun 7. PMID 31173437
- [Result] Pottier C, Ren Y, Perkerson RB 3rd, Baker M, Jenkins GD, van Blitterswijk M, DeJesus-Hernandez M, van Rooij JGJ, Murray ME, Christopher E, McDonnell SK, Fogarty Z, Batzler A, Tian S, Vicente CT, Matchett B, Karydas AM, Hsiung GR, Seelaar H, Mol MO, Finger EC, Graff C, Oijerstedt L, Neumann M, Heutink P, Synofzik M, Wilke C, Prudlo J, Rizzu P, Simon-Sanchez J, Edbauer D, Roeber S, Diehl-Schmid J, Evers BM, King A, Mesulam MM, Weintraub S, Geula C, Bieniek KF, Petrucelli L, Ahern GL, Reiman EM, Woodruff BK, Caselli RJ, Huey ED, Farlow MR, Grafman J, Mead S, Grinberg LT, Spina S, Grossman M, Irwin DJ, Lee EB, Suh E, Snowden J, Mann D, Ertekin-Taner N, Uitti RJ, Wszolek ZK, Josephs KA, Parisi JE, Knopman DS, Petersen RC, Hodges JR, Piguet O, Geier EG, Yokoyama JS, Rissman RA, Rogaeva E, Keith J, Zinman L, Tartaglia MC, Cairns NJ, Cruchaga C, Ghetti B, Kofler J, Lopez OL, Beach TG, Arzberger T, Herms J, Honig LS, Vonsattel JP, Halliday GM, Kwok JB, White CL 3rd, Gearing M, Glass J, Rollinson S, Pickering-Brown S, Rohrer JD, Trojanowski JQ, Van Deerlin V, Bigio EH, Troakes C, Al-Sarraj S, Asmann Y, Miller BL, Graff-Radford NR, Boeve BF, Seeley WW, Mackenzie IRA, van Swieten JC, Dickson DW, Biernacka JM, Rademakers R. Genome-wide analyses as part of the international FTLD-TDP whole-genome sequencing consortium reveals novel disease risk factors and increases support for immune dysfunction in FTLD. Acta Neuropathol. 2019 Jun;137(6):879-899. doi: 10.1007/s00401-019-01962-9. Epub 2019 Feb 9. PMID 30739198
- [Result] Staffaroni AM, Ljubenkov PA, Kornak J, Cobigo Y, Datta S, Marx G, Walters SM, Chiang K, Olney N, Elahi FM, Knopman DS, Dickerson BC, Boeve BF, Gorno-Tempini ML, Spina S, Grinberg LT, Seeley WW, Miller BL, Kramer JH, Boxer AL, Rosen HJ. Longitudinal multimodal imaging and clinical endpoints for frontotemporal dementia clinical trials. Brain. 2019 Feb 1;142(2):443-459. doi: 10.1093/brain/awy319. PMID 30698757
- [Result] Boeve BF, Rosen HJ. Multimodal imaging in familial FTLD: phenoconversion and planning for the future. Brain. 2019 Jan 1;142(1):8-11. doi: 10.1093/brain/awy314. PMID 30596906
- [Result] Toller G, Ranasinghe K, Cobigo Y, Staffaroni A, Appleby B, Brushaber D, Coppola G, Dickerson B, Domoto-Reilly K, Fields J, Fong J, Forsberg L, Ghoshal N, Graff-Radford N, Grossman M, Heuer H, Hsiung GY, Huey E, Irwin D, Kantarci K, Kaufer D, Kerwin D, Knopman D, Kornak J, Kramer J, Litvan I, Mackenzie I, Mendez M, Miller B, Rademakers R, Ramos E, Rascovsky K, Roberson E, Syrjanen J, Tartaglia C, Weintraub S, Boeve B, Boxer A, Rosen H, Rankin K; ARTFL/LEFFTDS Consortium. Revised Self-Monitoring Scale: A potential endpoint for frontotemporal dementia clinical trials. Neurology. 2020 Jun 2;94(22):e2384-e2395. doi: 10.1212/WNL.0000000000009451. Epub 2020 May 5. PMID 32371446
- [Result] Casaletto KB, Staffaroni AM, Wolf A, Appleby B, Brushaber D, Coppola G, Dickerson B, Domoto-Reilly K, Elahi FM, Fields J, Fong JC, Forsberg L, Ghoshal N, Graff-Radford N, Grossman M, Heuer HW, Hsiung GY, Huey ED, Irwin D, Kantarci K, Kaufer D, Kerwin D, Knopman D, Kornak J, Kramer JH, Litvan I, Mackenzie IR, Mendez M, Miller B, Rademakers R, Ramos EM, Rascovsky K, Roberson ED, Syrjanen JA, Tartaglia MC, Weintraub S, Boeve B, Boxer AL, Rosen H, Yaffe K; ARTFL/LEFFTDS Study. Active lifestyles moderate clinical outcomes in autosomal dominant frontotemporal degeneration. Alzheimers Dement. 2020 Jan;16(1):91-105. doi: 10.1002/alz.12001. PMID 31914227
- [Result] Kornak J, Fields J, Kremers W, Farmer S, Heuer HW, Forsberg L, Brushaber D, Rindels A, Dodge H, Weintraub S, Besser L, Appleby B, Bordelon Y, Bove J, Brannelly P, Caso C, Coppola G, Dever R, Dheel C, Dickerson B, Dickinson S, Dominguez S, Domoto-Reilly K, Faber K, Ferrall J, Fishman A, Fong J, Foroud T, Gavrilova R, Gearhart D, Ghazanfari B, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford N, Grant IM, Grossman M, Haley D, Hsiao J, Hsiung R, Huey ED, Irwin D, Jones D, Jones L, Kantarci K, Karydas A, Kaufer D, Kerwin D, Knopman D, Kraft R, Kramer J, Kukull W, Lapid M, Litvan I, Ljubenkov P, Lucente D, Lungu C, Mackenzie I, Maldonado M, Manoochehri M, McGinnis S, McKinley E, Mendez M, Miller B, Multani N, Onyike C, Padmanabhan J, Pantelyat A, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin K, Rascovsky K, Roberson ED, Rogalski-Miller E, Sengdy P, Shaw L, Staffaroni AM, Sutherland M, Syrjanen J, Tartaglia C, Tatton N, Taylor J, Toga A, Trojanowski J, Wang P, Wong B, Wszolek Z, Boeve B, Boxer A, Rosen H; ARTFL/LEFFTDS Consortium. Nonlinear Z-score modeling for improved detection of cognitive abnormality. Alzheimers Dement (Amst). 2019 Dec 5;11:797-808. doi: 10.1016/j.dadm.2019.08.003. eCollection 2019 Dec. PMID 31872042
- [Result] Boeve B, Bove J, Brannelly P, Brushaber D, Coppola G, Dever R, Dheel C, Dickerson B, Dickinson S, Faber K, Fields J, Fong J, Foroud T, Forsberg L, Gavrilova R, Gearhart D, Ghoshal N, Goldman J, Graff-Radford J, Graff-Radford N, Grossman M, Haley D, Heuer H, Hsiung GR, Huey E, Irwin D, Jones D, Jones L, Kantarci K, Karydas A, Knopman D, Kornak J, Kraft R, Kramer J, Kremers W, Kukull W, Lapid M, Lucente D, Mackenzie I, Manoochehri M, McGinnis S, Miller B, Pearlman R, Petrucelli L, Potter M, Rademakers R, Ramos EM, Rankin K, Rascovsky K, Sengdy P, Shaw L, Syrjanen J, Tatton N, Taylor J, Toga A, Trojanowski J, Weintraub S, Wong B, Wszolek Z, Boxer A, Rosen H; LEFFTDS Consortium. The longitudinal evaluation of familial frontotemporal dementia subjects protocol: Framework and methodology. Alzheimers Dement. 2020 Jan;16(1):22-36. doi: 10.1016/j.jalz.2019.06.4947. Epub 2020 Jan 6. PMID 31636026
- [Result] Miyagawa T, Brushaber D, Syrjanen J, Kremers W, Fields J, Forsberg LK, Heuer HW, Knopman D, Kornak J, Boxer A, Rosen H, Boeve B; ARTFL/LEFFTDS Consortium. Use of the CDR(R) plus NACC FTLD in mild FTLD: Data from the ARTFL/LEFFTDS consortium. Alzheimers Dement. 2020 Jan;16(1):79-90. doi: 10.1016/j.jalz.2019.05.013. Epub 2020 Jan 6. PMID 31477517
- [Derived] Tipton PW, Deutschlaender AB, Savica R, Heckman MG, Brushaber DE, Dickerson BC, Gavrilova RH, Geschwind DH, Ghoshal N, Graff-Radford J, Graff-Radford NR, Grossman M, Hsiung GR, Huey ED, Irwin DJ, Jones DT, Knopman DS, McGinnis SM, Rademakers R, Ramos EM, Forsberg LK, Heuer HW, Onyike C, Tartaglia C, Domoto-Reilly K, Roberson ED, Mendez MF, Litvan I, Appleby BS, Grant I, Kaufer D, Boxer AL, Rosen HJ, Boeve BF, Wszolek ZK; ALLFTD Consortium. Differences in Motor Features of C9orf72, MAPT, or GRN Variant Carriers With Familial Frontotemporal Lobar Degeneration. Neurology. 2022 Sep 13;99(11):e1154-e1167. doi: 10.1212/WNL.0000000000200860. Epub 2022 Jul 5. PMID 35790423
- [Derived] Gendron TF, Heckman MG, White LJ, Veire AM, Pedraza O, Burch AR, Bozoki AC, Dickerson BC, Domoto-Reilly K, Foroud T, Forsberg LK, Galasko DR, Ghoshal N, Graff-Radford NR, Grossman M, Heuer HW, Huey ED, Hsiung GR, Irwin DJ, Kaufer DI, Leger GC, Litvan I, Masdeu JC, Mendez MF, Onyike CU, Pascual B, Ritter A, Roberson ED, Rojas JC, Tartaglia MC, Wszolek ZK, Rosen H, Boeve BF, Boxer AL; ALLFTD consortium; Petrucelli L. Comprehensive cross-sectional and longitudinal analyses of plasma neurofilament light across FTD spectrum disorders. Cell Rep Med. 2022 Apr 19;3(4):100607. doi: 10.1016/j.xcrm.2022.100607. eCollection 2022 Apr 19. PMID 35492244
- [Derived] Rojas JC, Wang P, Staffaroni AM, Heller C, Cobigo Y, Wolf A, Goh SM, Ljubenkov PA, Heuer HW, Fong JC, Taylor JB, Veras E, Song L, Jeromin A, Hanlon D, Yu L, Khinikar A, Sivasankaran R, Kieloch A, Valentin MA, Karydas AM, Mitic LL, Pearlman R, Kornak J, Kramer JH, Miller BL, Kantarci K, Knopman DS, Graff-Radford N, Petrucelli L, Rademakers R, Irwin DJ, Grossman M, Ramos EM, Coppola G, Mendez MF, Bordelon Y, Dickerson BC, Ghoshal N, Huey ED, Mackenzie IR, Appleby BS, Domoto-Reilly K, Hsiung GR, Toga AW, Weintraub S, Kaufer DI, Kerwin D, Litvan I, Onyike CU, Pantelyat A, Roberson ED, Tartaglia MC, Foroud T, Chen W, Czerkowicz J, Graham DL, van Swieten JC, Borroni B, Sanchez-Valle R, Moreno F, Laforce R, Graff C, Synofzik M, Galimberti D, Rowe JB, Masellis M, Finger E, Vandenberghe R, de Mendonca A, Tagliavini F, Santana I, Ducharme S, Butler CR, Gerhard A, Levin J, Danek A, Otto M, Sorbi S, Cash DM, Convery RS, Bocchetta M, Foiani M, Greaves CV, Peakman G, Russell L, Swift I, Todd E, Rohrer JD, Boeve BF, Rosen HJ, Boxer AL; ALLFTD and GENFI consortia. Plasma Neurofilament Light for Prediction of Disease Progression in Familial Frontotemporal Lobar Degeneration. Neurology. 2021 May 4;96(18):e2296-e2312. doi: 10.1212/WNL.0000000000011848. Epub 2021 Apr 7. PMID 33827960
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials
- See also: UCSF Research Trials — https://memory.ucsf.edu/research-trials/research